CLINICAL TRIAL: NCT06422195
Title: Does the Dynamic Needle Tip Positioning Modification Technique in Short Axis Approach (DNTP - SA) Provides a Faster Ultrasound-guided Arterial Cannulation Than Long Axis (LA) Approach: A Prospective Randomized Controlled Study
Brief Title: Dynamic Needle Tip Positioning Modification Technique in Short Axis Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Maram Ibrahim Elmazny, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 36197/12/22
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Dynamic Needle Tip Positioning; Short Axis; Arterial Cannulation; Long Axis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Needle Tip Positioning Technique in Short Axis Approach (DNTP - SA) (Experimental): Ultrasound guided radial artery cannulation by Dynamic Needle Tip Positioning Technique in Short Axis Approach (DNTP - SA) will be performed by an experienced anesthesiologist who has no subsequent role in the study. The ultrasound transducer is oriented transversely to the radial artery at the wrist, and the vessel appears as a circular anechoic structure in the ultrasound screen with gradual advancing of the needle till reaching the radial artery. Meanwhile, the ultrasound probe is being moved proximally in advance of the needle tip until it disappears from the ultrasound image. The cannula then advanced in the direction of the artery.
  Interventions: Other: Dynamic Needle Tip Positioning Technique in Short Axis Approach (DNTP - SA)
- Long Axis Approach (LA) (Active Comparator): Ultrasound guided radial artery cannulation in Long Axis Approach (LA) will be performed by an experienced anesthesiologist who has no subsequent role in the study. In the LA-IP approach, an ultrasound probe is placed parallel to the radial artery and the artery appears as a tubular anechoic structure in ultrasound.
  Interventions: Other: Long Axis Approach (LA)

INTERVENTIONS:
Other: Dynamic Needle Tip Positioning Technique in Short Axis Approach (DNTP - SA) — Ultrasound guided radial artery cannulation by Dynamic Needle Tip Positioning Technique in Short Axis Approach (DNTP - SA) will be performed by an experienced anesthesiologist who has no subsequent role in the study. The ultrasound transducer is oriented transversely to the radial artery at the wrist, and the vessel appears as a circular anechoic structure in the ultrasound screen with gradual advancing of the needle till reaching the radial artery. Meanwhile, the ultrasound probe is being moved proximally in advance of the needle tip until it disappears from the ultrasound image. The cannula then advanced in the direction of the artery.
  Arms: Dynamic Needle Tip Positioning Technique in Short Axis Approach (DNTP - SA)
Other: Long Axis Approach (LA) — Ultrasound guided radial artery cannulation in Long Axis Approach (LA) will be performed by an experienced anesthesiologist who has no subsequent role in the study. In the LA-IP approach, an ultrasound probe is placed parallel to the radial artery and the artery appears as a tubular anechoic structure in ultrasound.
  Arms: Long Axis Approach (LA)

SUMMARY:
The aim of the present study is to compare between Dynamic Needle Tip Positioning Modification Technique in Short Axis Approach (DNTP - SA) and Long Axis (LA) Approach for Ultrasound-guided Arterial Cannulation as regard time to successful arterial cannula insertion as well as the success rate in the first trial of insertion, number of attempts till successful arterial line placemen, complications, and operators' satisfaction.

DETAILED DESCRIPTION:
Intraoperative Arterial cannulation is recently frequently required especially in high-risk patients or patients with expected major fluid shift.

The most common site for arterial cannulation is the radial artery because of ease of accessibility, dual blood supply to the hand via the ulnar artery, and a low rate of complications. Complications from arterial cannulation include thrombosis, hematoma formation, edema and vasospasm.

Two approaches are basically identified for ultrasound-guided radial artery cannulation, i.e., short-axis out-of-plane (SA-OOP) and long-axis in-plane (LA-IP) techniques.

The dynamic needle tip positioning (DNTP) technique uses the short-axis view of the radial artery with gradual advancing of the needle till reaching the radial artery. Meanwhile, the ultrasound probe is being moved proximally in advance of the needle tip until it disappears from the ultrasound image. The cannula then advanced in the direction of the artery

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years.
* Both sexes.
* American Society of Anesthesiologists physical status II-IV.
* Patients scheduled for elective surgery procedure that requires the use of invasive arterial pressure monitoring, as determined by the attending anesthesiologist.

Exclusion Criteria:

* Emergency patients or with Hemodynamic instability.
* Patients who have cellulitis or infection at the site of insertion.
* Patients with a positive modified Allen test.
* Raynaud disease or any Peripheral vascular disease.
* Patients with Multiple previous radial artery interventional therapies in the previous 30 days.
* Patients scheduled for Surgery at site of insertion like forearm flap.
* Refusal to participate by the patient.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2024-05-19 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Time to achieve successful cannulation | Immediately after catheterization
  Time to achieve successful cannulation will be measured from initial skin puncture until the catheter is placed into the radial artery.

SECONDARY OUTCOMES:
The success rate | Immediately after catheterization
  The success rate in the first trial of insertion between the two different approaches will be assessed.
Number of attempts till successful arterial cannula insertion | Immediately after catheterization
  Number of attempts till successful arterial cannula insertion will be recorded.
Incidence of complications | 24 hours postoperatively
  Complications including edema, hematoma, vasospasm, ischemia, thrombosis and nerve injury will be recorded.
Operators' satisfaction | Immediately after catheterization
  Operators' satisfaction (Level of operators' satisfaction will be assessed with a Scale from 1-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

REFERENCES:
- [Derived] Elmazny MI, Ahmed S, Afifi S. Dynamic needle tip positioning in short-axis versus long-axis ultrasound-guided arterial cannulation: a randomised controlled trial. BMC Anesthesiol. 2025 Nov 14;25(1):561. doi: 10.1186/s12871-025-03413-3. PMID 41239242